CLINICAL TRIAL: NCT02322073
Title: Inflammation and Obesity-associated Disease
Acronym: Adipos2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 682-14
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Obesity; Inflammation; Kidney Disease; Liver Disease; Metabolic Syndrome; Cardiometabolic Syndrome; Fibrosis
MeSH Terms: conditions — Obesity; Inflammation; Kidney Diseases; Liver Diseases; Metabolic Syndrome; Fibrosis | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lean healthy controls: Healthy controls with BMI 18.5-24.9 Laparoscopic surgery eg cholecystectomy, fundoplication or Heller myotomy and fundoplication or laparoscopic hernia repair.
  Interventions: Procedure: Laparoscopic surgery
- Obese: Obese BMI 35-55 Laparoscopic Roux-en-Y gastric bypass or Sleeve gastrectomy Phenotype according to cardiometabolic status

INTERVENTIONS:
Procedure: Laparoscopic surgery — Roux-en-Y gastric bypass or other benign laparoscopic surgery
  Groups: Lean healthy controls

SUMMARY:
Visceral obesity and adipose inflammation is considered a driving force of obesity-related systemic disease, e.g. cardiometabolic disease, liver cirrhosis and chronic kidney disease (CKD). Inflammatory resolution is actively regulated by specialized pro-resolving mediators (SPMs), including the endogenous eicosanoid LXA4. Impairment of SPMs may underlie development of obesity-related pathology.We hypothesize that obese patients who develop obesity-related disease do so because they suffer from impaired endogenous production of pro-resolving lipids. This will result in aggravated adipose inflammation and fibrosis, which contribute to the systemic pathologies. We thus wish to investigate adipose inflammation and the pro-resolving lipid profile of obese subjects with and without obesity associated metabolic disease. We also aim to investigate whether LXA4, LXB4 and other anti-inflammatory agents (such as AICAR) can alter the phenotype of human adipose macrophages in ex vivo tissue culture. We also investigate basic pathways in inflammatory regulation and obesity related cardiometabolic disease.

ELIGIBILITY:
Inclusion Criteria:

* Obese BMI 35-55 kg/m2
* Lean BMI 18.5-24.9

Exclusion Criteria:

* Medical treatment with NSAIDs, corticosteroid treatment, immune-suppressants.
* Other: smoking, alcohol abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese individuals planned for Roux-en-Y gastric bypass or Sleeve gastrectomy surgery and lean healthy controls planned for elective benign laparoscopic surgery.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-12-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Inflammatory status | One year
  inflammatory status vs cardiometabolic disease and tissue fibrosis

CONTACTS AND LOCATIONS:
Locations (1):
- Sahglrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Borgeson E, Wallenius V, Syed GH, Darshi M, Lantero Rodriguez J, Biorserud C, Ragnmark Ek M, Bjorklund P, Quiding-Jarbrink M, Fandriks L, Godson C, Sharma K. AICAR ameliorates high-fat diet-associated pathophysiology in mouse and ex vivo models, independent of adiponectin. Diabetologia. 2017 Apr;60(4):729-739. doi: 10.1007/s00125-017-4211-9. Epub 2017 Feb 10. PMID 28188334